CLINICAL TRIAL: NCT06816511
Title: Preliminary Explorative Study of Magnetic Resonance-Guided Focused Ultrasound Surgery in Refractory Obsessive-Compulsive Disorder Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202307078DIND
Record Dates: First submitted 2024-12-26; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: Magnetic Resonance-Guided Focused Ultrasound; Refractory Obsessive-Compulsive Disorder; anterior limb of the internal capsule; functional magnetic resonance imaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Procedure: magnetic resonance-guided focused ultrasound surgery, MRgFUS

INTERVENTIONS:
Procedure: magnetic resonance-guided focused ultrasound surgery, MRgFUS — Magnetic Resonance-Guided Focused Ultrasound Surgery The clinical symptoms, brain imaging, and cognitive function status were followed up for 2 years before and after surgery.

SUMMARY:
The goal of this clinical trial is to evaluate If magnetic resonance-guided focused ultrasound works to treat refractory obsessive-compulsive disorder in adults. The main questions it aims to answer are:

* What effectiveness does the magnetic resonance-guided focused ultrasound bring to the participants during study period?
* What side effects do the participant have when treated with magnetic resonance-guide focused ultrasound?

Participants will:

* Finish scales to evaluate participants' level of cognitive function, depression and Compulsiveness.
* Receive the treatment of magnetic resonance-guided focused ultrasound
* Take the fMRI brain scanning before and after the treatment
* Recovering

ELIGIBILITY:
Inclusion Criteria:

* For 30 days before enrollment, the type and dosage of primary OCD medications (including antidepressants and adjunctive medications such as antipsychotics and tricyclic antidepressants) remain unchanged. However, other symptom-relief medications, such as anti-anxiety drugs, are not restricted.
* Diagnosed by a psychiatrist through a diagnostic interview, meeting the criteria for OCD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) for at least five years; and scoring above 28 on the Chinese version of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS).
* OCD symptoms show limited improvement with existing treatments, classified as refractory according to the OCD Clinical Practice Review Task Force of the Anxiety & Depression Association of America (ADAA):

  i. Received treatment with at least three different antidepressants at adequate doses and durations.

ii. Received treatment with at least two of the following medications for over a month each: antipsychotics, clonazepam, lithium, buspirone.

iii. Underwent appropriate cognitive-behavioral therapy with exposure and response prevention (EX/RP) for at least 20 sessions.

* Able to comply with focused ultrasound-related operational instructions (device: ExAblate MRgFUS). During the procedure, participants must be able to communicate with the physician and express their sensory experiences (general anesthesia is not required).
* After explanation by a psychiatrist and neurosurgeon, participants provide informed consent and can comply with the research process and related guidance. During the trial, participants must be able to independently press the stop-ultrasound button.

Exclusion Criteria:

- Major and Potential Physical Conditions That May Affect the Treatment Process: i. Cardiovascular or hemodynamic abnormalities, such as heart failure, arrhythmias, tachycardia or bradycardia (>100 bpm, <60 bpm), abnormal systolic blood pressure (>180 mmHg, <90 mmHg), abnormal diastolic blood pressure (>180 mmHg), and severe hypertension uncontrolled by medication (diastolic blood pressure >100 mmHg after stable medication use). Additionally, those who have taken medications affecting autonomic regulation and potentially impacting vital sign stability within six months before treatment (however, antidepressants and antipsychotics taken for mental illness are not included).

ii. Platelet or coagulation disorders or currently taking anticoagulant medications (e.g., Warfarin, Avastin).

iii. Renal dysfunction (eGFR < 30ml/min/1.73 m²) or currently undergoing hemodialysis.

iv. Severe infections. v. Immunocompromised individuals. vi. History of intracranial hemorrhage, intracranial aneurysm, cerebrovascular events within six months, or brain tumors.

vii. Neurological disorders: stroke, epilepsy, suspected increased intracranial pressure (IICP), Parkinson's disease and related disorders (Multisystem atrophy, Progressive supranuclear palsy, Dementia with Lewy bodies, Alzheimer's disease).

viii. Other clinically assessed physical conditions that may pose significant risks to bodily functions and life during the treatment process.

* Patients deemed unsuitable for magnetic resonance-guided focused ultrasound after evaluation, including those with low skull density ratio (<0.4), intracranial implants, or structures that cannot avoid energy-absorbing or sensitive tissues in the ultrasound path (e.g., previous brain shunt sites, surgical metal clips, significant calcification, extensive scarring, or any rigid implants). (Pre-treatment evaluation will include a head CT scan to calculate the skull density ratio (SDR) to determine suitability for focused ultrasound treatment; a low SDR may affect the efficiency of the treatment and increase side effects, making the patient unsuitable for treatment.)
* Bilateral structural abnormalities in the anterior limb of the internal capsule (ALIC).
* Contraindications to MRI or its contrast agents, or incompatible metal implants in the body.
* Inability to comply with treatment instructions, lack of behavioral capacity, or lack of treatment motivation.
* Major psychiatric comorbidities: schizophrenia spectrum disorders, acute episodes, bipolar disorder, acute episodes, severe dementia, unresolved alcohol or substance abuse, recent suicidal ideation or plans.
* Pregnancy or breastfeeding.
* Scalp atrophy or difficulty healing scalp wounds.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | For two years after the surgery

SECONDARY OUTCOMES:
Clinical Symptoms | For two years after the surgery
  Chinese version of the Yale-Brown Obsessive-Compulsive Scale, Chinese version of the Montgomery Depression Scale, Chinese version of the Hamilton Anxiety Scale.
Structural Brain Imaging | For two years after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided